CLINICAL TRIAL: NCT03110406
Title: Effects of Whole-body Vibration Training on the Heart Rate Variability Cardiac in Kidney Transplantation: a Randomized Controlled Trial
Brief Title: Effects of Whole-body Vibration Training on the Heart Rate Variability Cardiac in Kidney Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, TUIRA OLIVEIRA MAIA, Master, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TUIRAMAIA
Record Dates: First submitted 2017-03-22; First posted 2017-04-12 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Renal Transplant Recipients
Keywords: renal transplant recipients; exercise; heart rate variability; Cardiovascular mortality
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Intervention group and control group
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- whole-body vibration (Experimental): The whole-body vibration training will be performed with the patients in the static position, feet apart at 20 cm, semi-squat with knees at 15º flexion and upper limbs slightly flexed and supported on the platform. The exercises will be performed, in the first two weeks, for 10 minutes consisting of 60 seconds of low intensity with 30 seconds of rest standing in the anatomical position. From the second week to the end of the twelfth week (24 sessions) will be performed 15 minutes corresponding being 60 seconds of high intensity interspersed with 30 seconds of rest standing in the anatomical position. In the second month, the patient should be well adapted to the stimuli of the platform keeping the frequency of 35Hz and the amplitude 4mm. °
  Interventions: Other: whole-body vibration training
- Simulated whole-body vibration (Sham Comparator): The simulated whole-body vibration training will be performed with the patients in the static position, feet apart at 20 cm, in semi-squat with knees at 15º of flexion and upper limbs slightly flexed and supported on the platform that presents a motor that simulates the noise of the platform But does not produce any therapeutic effect
  Interventions: Other: whole-body vibration training

INTERVENTIONS:
Other: whole-body vibration training — Training on the Vibrating platform will be performed with the patients in the static position.The exercises will be performed in the first two weeks for 10 minutes consisting of 60 seconds of low intensity and 30 seconds of standing rest in the anatomical position. From the second week to the end of the twelfth week (24 sessions) will be performed 15 minutes corresponding being 60 seconds of high intensity interspersed with 30 seconds of rest standing in the anatomical position. In the second month, the patient should be well adapted to the stimuli of the platform keeping the frequency of 35Hz and the amplitude 4mm. Monitoring of blood pressure, heart rate and peripheral oxygen saturation should be done every 5 minutes.

SUMMARY:
Introduction: Renal transplantation represents the therapeutic mode with more durable treatment, greater cost-effectiveness, survival benefits and quality of life of the patients, however, with high cardiovascular mortality.

Objectives: To evaluate the acute and chronic effects on heart rate variability and the impact of chronic kidney disease on cardiorespiratory fitness in renal transplant recipients following a full-body Vibration training program.

Methods: It will be a blinded randomized clinical trial (patient, evaluator and statistician), controlled and endowed with secrecy of allocation, to be performed in the Cardiopulmonary Physiotherapy Laboratory of the Physiotherapy Department of the Federal University of Pernambuco. Renal transplant recipients will be recruited at the Nephrology outpatient clinic of the Hospital das Clínicas de Pernambuco, according to the following inclusion criteria: age between 18 and 59 years, who underwent transplantation at least one year before and present a stable transplant function through the level Of creatinine

DETAILED DESCRIPTION:
It will be a blinded randomized clinical trial (patient, evaluator and statistician), controlled and endowed with secrecy of allocation, to be performed in the Cardiopulmonary Physiotherapy Laboratory of the Physiotherapy Department of the Federal University of Pernambuco. Renal transplant recipients will be recruited at the Nephrology outpatient clinic of the Hospital das Clínicas de Pernambuco, according to the inclusion criteria

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 59 years
* who underwent transplantation at least one year before
* present a stable transplantation function through the creatinine level <1.8 mg / dL
* No drug use with ability to modify the autonomic nervous system, such as sympatholytic drugs

Exclusion Criteria:

* unstable hypertension;
* Amyloidosis;
* Congestive heart failure, recent myocardial infarction, unstable angina;
* Musculoskeletal abnormality that impairs the performance of the exercises;
* Have a metal implant or cardiac pacemaker.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-03-10 (Actual); Primary Completion 2017-09-30 (Estimated); Study Completion 2018-03-10 (Estimated)

PRIMARY OUTCOMES:
heart rate variability | three months
  Heart rate variability will be assessed through holter

SECONDARY OUTCOMES:
Oxygen consumption | three months
  Oxygen consumption will be assessed through exercise test

CONTACTS AND LOCATIONS:
Overall Officials: TUIRA O M, Principal Investigator — UFPE
Locations (1):
- Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No